CLINICAL TRIAL: NCT01906827
Title: P-wave Duration and Dispersion in Intrahepatic Cholestasis of Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Ayse Kirbas, ayse kirbas, Zekai Tahir Burak Women's Health Research and Education Hospital
Other Study IDs: zekai tahir burak- p wave
Record Dates: First submitted 2013-07-20; First posted 2013-07-24 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2013-07

CONDITIONS: Intrahepatic Cholestasis of Pregnancy; Arrhythmia
Keywords: cholestasis; pregnancy; p wave dispersion; arrhythmia
MeSH Terms: conditions — Intrahepatic Cholestasis of Pregnancy; Arrhythmias, Cardiac; Cholestasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pregnant with ICP: pregnant with ICP

SUMMARY:
The bile acids has been demonstrated to cause arrhythmia and abnormal calcium dynamics in cultured neonatal rat cardiomyocytes. Bile acids may alter maternal cardiomyocyte function like fetus.Increased P-wave duration and P-wave dispersion have been reported in various clinical settings. The investigators hypothesized that PWD and p wave duration may affect in pregnancy with ICP.

DETAILED DESCRIPTION:
Intrahepatic cholestasis of pregnancy (ICP) is a pregnancy-specific liver disease. The most frequent laboratory abnormality is elevation of serum bile acid levels in ICP.

Bile acids increases both maternal and fetal circulation in ICP. The bile acids has been demonstrated to cause arrhythmia and abnormal calcium dynamics in cultured neonatal rat cardiomyocytes. Raised maternal bile acid levels have been associated with fetal distress and arrhytmia in fetus.

P-wave dispersion (PWD) is defined as the difference between the maximum and the minimum P-wave durations measured on a 12-lead surface electrocardiogram (ECG). Increased P-wave duration and PWD have been reported in various clinical settings, including atrial flutter, coronary artery disease, hypertension, rheumatic mitral stenosis, mitral annular calcification, obstructive sleep apnea, and obesity.

So the investigators think that bile acids may alter maternal cardiomyocyte function as fetus. The investigators hypothesized that PWD and p wave duration may affect in pregnancy with ICP.

The aim of this study is to investigate maternal P-wave duration and dispersion changes in pregnant women with intrahepatic cholestasis of pregnancy .

ELIGIBILITY:
Inclusion Criteria:

- Pregnants who with ICP

Exclusion Criteria:

* Chronic liver disease
* Disease during current pregnancy
* Multiple pregnancies

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The pregnant women with intrahepatic cholestasis who admitted our clinic
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-05 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
change in the range of P-wave Duration and Dispersion | one year
  A 12-lead surface ECG will obtain for all pregnants with icp in the supine position after a rest period of 10 minutes. Two consecutive cycles will record at a speed of 50 mm/sec and with an amplitude of 10mm/mV. All ECGs will examine by a designated cardiologist blinded to patient details. To improve accuracy, measurements will made using calipers and magnifying lens. Only participants with normal sinus rhythm on ECG will include in the final analysis

CONTACTS AND LOCATIONS:
Overall Officials: ayse kirbas, md, Principal Investigator — Zekai Tahir Burak Women's Health Research and Education Hospital; ozgur kirbas, md, Principal Investigator — Yuksek Ihtisas Hospital
Locations (1):
- Zekai Tahir Burak Maternity Teaching Hospital, Ankara, Turkey (Türkiye)